CLINICAL TRIAL: NCT05520788
Title: Ambispective Cohort Study of Precision Medicine for Primary Hepatobiliary Cancer Based on Next-generation Sequencing
Acronym: CCGLC-006
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ze-yang Ding, MD, Prof., Tongji Hospital
Other Study IDs: TJ-IRB20220129
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer
Keywords: Liver Neoplasms; Biliary Tract Neoplasms; NGS
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The samples, both tissue(s) and blood of patients should be provided for the High-Throughput Sequencing test before screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Precise medicine: All patients should accept next-generation sequencing (NGS) test before treatment.
  Interventions: Genetic: precise medicine

INTERVENTIONS:
Genetic: precise medicine — During screening stage, all patients should accept next-generation sequencing (NGS) test.

SUMMARY:
Exploring the precise medicine of patients with primary hepatobiliary cancer. And evaluate the efficacy and safety of individualized treatment regimens for primary hepatobiliary cancer based on next-generation sequencing.

DETAILED DESCRIPTION:
The purpose of this study is to explore the precise treatment in hepatobiliary cancer patients and evaluate drug efficacy, progression free and overall survival. This trial study is based on genetic tests, then therapeutic target drugs are administered according to the genetic test reports. Patients with genetic abnormalities (such as mutations, amplifications, or translocations) may benefit from precise treatment which targets particular genetic abnormality. The identifications of these genetic abnormalities may help treat hepatobiliary cancer patients.

The genetic tests are performed for the eligible subjects in this study, then therapeutic target drugs are administered according to the genetic test reports. While the precise treatments, follow-ups are conducted to evaluate the efficacy and safety of the target drugs for the subjects, until the overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65, male or female.
2. Radiologically and pathologically confirmed as hepatobiliary cancers with stage IV.
3. Palliative care as the preferred.
4. The result of next-generation sequencing (NGS) test show the patient has gene mutation and also can be treated by the right commercial products that have been approved by the China Food and Drug Administration (CFDA) or the Food and Drug Administration (FDA).
5. ECOG performance status 0-2.
6. Life expectancy ≥3 months.
7. Agree to sign informed consent form.

Exclusion Criteria:

1. Hepatobiliary cancer patient with stageI-III, or with any of the following items will not be eligible for screening. Such as, suitable for the treatment of radical resection, radical resection but evaluation unmeasurable.
2. The result of NGS test show the patient has no gene mutation, or has gene mutation but no medicine.
3. ECOG performance status ≥ 3.
4. Female patients who are pregnant or not using a contraceptive method of birth control.
5. History or presence of serious cardiovascular or cerebrovascular abnormalities.
6. Abnormalities of the hepatic or renal functions, such as jaundice, ascites, bilirubin ≥ 1.5×ULN, alkaline phosphatase ≥ 3×ULN, persistent protein urine≥ grade 3 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0), creatinine ratio > 3.5g/24 hours, renal failure.
7. Persistent infection > grade 2 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0).
8. Patient has underwent a major operation 4 weeks prior to screening or has not yet recovered from the operation.
9. Patient with epilepsy, known or untreated brain metastases.
10. The presence of wounds, ulcers or fractures that can not be healed, or with a past history of transplantation.
11. The presence of bleeding events ≥grade 3 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0) , present evidence or past history of coagulation dysfunction disorders.
12. Known human immunodeficiency virus (HIV) infection history.
13. Patient with drug abuse or unstable compliance.
14. The presence of unresolved toxicity caused by any previous treatment/operation > grade 1 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0), except alopecia, anemia or hypothyroidism).
15. Investigator consider that the patient should not be enrolled in this study by careful assessment.
16. The subjects participate in any other clinical trial in the meantime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed primary hepatobiliary cancer in Tongji Hospital, Wuhan with results of NGS tests.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From treatment initiation for advanced or metastatic HCC to the first date of disease progression for any cause up to 2 year
  Time of progression will be obtained by telephone interview or medical treatment records.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Include all-cause death of patients in this study.
Objective response rates (ORR) | From treatment initiation to CR or PR, up to 2 years
  Percentage of patients whose tumors have a complete or partial response to treatment.
Disease Control Rate (DCR) | From treatment initiation to SD, CR or PR, up to 2 years
  The proportion of patients who had either stable disease (SD) for ≥ 6 months, a CR or PR after initiation of treatment for HCC
Duration of Response (DOR) | From treatment initiation to PD, up to 2 years
  duration from the first assessment of the tumor was CR or PR to the time that the first assessment for PD or date of death from any cause
Adverse Drug Reaction (ADR)/Adverse Event (AE) | Through study completion, an average of 2 years.
  Patients with treatment-related adverse events as assessed by CTCAE v4.0.
Quality of Life (QoL) after treatment | Through study completion, an average of 2 years.
  The life quality of every subject will be assessed every 3 months according to the FACT-Hep questionnaire, which assesses generic HRQL concerns and disease-specific issues.

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, Study Chair — Tongji Hospital; Zeyang Ding, Principal Investigator — Tongji Hospital
Locations (1):
- Hepatic Surgery Center, Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The data have the gene mutations information of patients.